CLINICAL TRIAL: NCT02043262
Title: Evaluating Reablement for Home-dwelling Elderly in a Norwegian Municipality
Brief Title: The Effectiveness of Reablement in Home Dwelling Older Adults. A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frode F. Jacobsen (Other)
Collaborators: University of Bergen (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor-Investigator, Frode F. Jacobsen, Professor, Bergen University College
Organization: Bergen University College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/295
Record Dates: First submitted 2012-11-20; First posted 2014-01-23 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Physical Disability
Keywords: Elderly; Home-based rehabilitation; Activities of daily living; Restorative care; Reablement; Everyday rehabilitation
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reablement (Experimental): Reablement is an intensive, multidisciplinary, client-centered, home-based type of rehabilitation, where ordinary activities of daily living are used for rehabilitative purposes. It is a rehabilitation alternative that may be offered to older adults, although there is no lower age limit. An occupational therapist and physical therapist, or nurse, constitutes the key personal, while home helpers, assistants and others with lower education, are the ones who work rehabilitative with the older person on a daily basis focusing on self-help.
  Interventions: Behavioral: Reablement
- Standard treatment (Active Comparator): This arm consists of the standard treatment home-dwelling elderly persons receive when applying for home-based help. Some elderly may receive home-based nursing or home help services assisting them in daily activities, while others may receive occupational therapy or physical therapy measures for rehabilitative purposes.
  Interventions: Behavioral: Standard treatment

INTERVENTIONS:
Behavioral: Reablement — The intervention deals with improving function in daily activities the person defines as important in the areas of self-care, productivity and leisure.
  Other Names: Hverdagsrehabilitering; Hemrehabilitering; Re-ablement; Restorative care
  Arms: Reablement
Behavioral: Standard treatment — The control intervention is standard home-based treatment/care in Norway.
  Other Names: Usual care; Treatment as usual
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to determine whether a special kind of rehabilitation offered to home-dwelling older adults is effective with regards to functional ability and municipal costs.

DETAILED DESCRIPTION:
Early detection of functional decline among home dwelling older adults and immediate onset of rehabilitation, can improve function, and reduce or delay need for home-based assistance and nursing home placement. Towards year 2050 there will be a significant increase in number of elderly persons in Norway, with an urgent need for new models for early intervention and rehabilitation in order to give service to a larger amount of elderly persons. Reablement is a new and promising rehabilitation model which many Norwegian municipalities are implementing in order to meet current and future needs for municipal home-based services. However, very little research has been conducted regarding the effectiveness of this intervention. This study aims at assessing the effectiveness of reablement in terms of daily functioning and economic costs compared to standard home-based treatment and care.

The study will be conducted in the municipality of Voss in Western Norway, a municipality with only 14000 inhabitants. It is a double-blinded, block-randomized controlled intervention trial, recruiting home-dwelling older adults with an initial functional decline in daily activities. The intervention is intensive, multidisciplinary, home-based rehabilitation given by home-trainers, under supervision from an occupational therapist or a physiotherapist. The control intervention is standard home-based treatment and care.

Thirty participants will be recruited in each arm of the study. The participants will be assessed at baseline, and at 3-, and 9 months follow-up. Primary outcomes will be participation, activity, and municipal expenditures. Costs are generated by the working hours of the different professions. Hence, there will be a daily registration of the working hours different health care professions spend in the private homes of the participants.

Power calculations based on study with a similar target group using the instrument Canadian Occupational Performance Measure, estimate a need for only 21 participants in each group due to the longitudinal design. However, in order to account for possibilities of frailer target group or a large drop out rate (40 %), a total number of 30 participants in each group will be tried recruited. Data analyses will be performed according to intention to treat. The working hour data is panel data and will be analyzed accordingly; a random or a mixed effect regression model will be employed. Also, descriptive statistics and simpler tests will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Home-dwelling person
* Applicant of home-based services
* Above 18 years old
* Functional decline in at least one activity
* Able to understand written and oral Norwegian

Exclusion Criteria:

* Cognitive disability
* Terminal ill
* Being assessed as needing nursing home placement
* Being assessed as needing institution-based rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline
  Activity and participation will be measured using Canadian Occupational Performance Measure (COPM) The COPM is a measure of a client's self-perception of occupational performance in the areas of self-care, productivity and leisure. Outcome measures for the COPM are: the client's most important problems in occupational performance and a total score of performance and a total score of satisfaction for these problems.
Canadian Occupational Performance Measure | 3 months
  Activity and participation will be measured using Canadian Occupational Performance Measure (COPM) The COPM is a measure of a client's self-perception of occupational performance in the areas of self-care, productivity and leisure.
Canadian Occupational Performance Measure | 9 months
  Activity and participation will be measured using Canadian Occupational Performance Measure (COPM) The COPM is a measure of a client's self-perception of occupational performance in the areas of self-care, productivity and leisure.

SECONDARY OUTCOMES:
Expenditure | Daily from baseline to 9 months.
  Municipal expenditures will be recorded daily for nine months. Costs will be recorded in accordance with the operating hours of the different health care professions in the private homes of the participants. The control group will be assessed for amount of municipal home-based help at 15 months follow-up.
Expenditure | 15 months follow-up
  The control group will be assessed for amount of municipal home-based help at 15 months follow-up.

OTHER OUTCOMES:
Timed Up and Go | Baseline
  Mobility will be measured using "The Timed Up and Go" (TUG). This is a simple, clinical performance-based measure of lower extremity function, mobility and fall risk. Normative data exists.
COOP/Wonka | Baseline
  COOP/Wonka is a generic patient oriented instrument covering the domains of physical fitness, feelings, daily activities, social activities, change in health and overall health.
Dynamometer | Basline
  Hand strength will be measured with a hydraulic hand dynamometer. Normative grip strength data exists.
Timed Up and Go | 3 months
  Mobility will be measured using "The Timed Up and Go" (TUG). This is a simple, clinical performance-based measure of lower extremity function, mobility and fall risk.
Timed Up and Go | 9 months
  Mobility will be measured using "The Timed Up and Go" (TUG). This is a simple, clinical performance-based measure of lower extremity function, mobility and fall risk.
COOP/Wonka | 3 months
  COOP/Wonka is a generic patient oriented instrument covering the domains of physical fitness, feelings, daily activities, social activities, change in health and overall health.
COOP/Wonka | 9 months
  COOP/Wonka is a generic patient oriented instrument covering the domains of physical fitness, feelings, daily activities, social activities, change in health and overall health.
Dynamometer | 3 months
  Hand strength will be measured with a hydraulic hand dynamometer.
Dynamometer | 9 months
  Hand strength will be measured with a hydraulic hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Frode Fa Jacobsen, PhD, Study Chair — Bergen University College
Locations (2):
- Norway (2):
  - Bergen University College, Bergen
  - Municpality of Voss, Bergen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tuntland H, Aaslund MK, Espehaug B, Forland O, Kjeken I. Reablement in community-dwelling older adults: a randomised controlled trial. BMC Geriatr. 2015 Nov 4;15:145. doi: 10.1186/s12877-015-0142-9. PMID 26537789
- [Derived] Tuntland H, Espehaug B, Forland O, Hole AD, Kjerstad E, Kjeken I. Reablement in community-dwelling adults: study protocol for a randomised controlled trial. BMC Geriatr. 2014 Dec 18;14:139. doi: 10.1186/1471-2318-14-139. PMID 25519828
- See also: Published randomised controlled trial — https://www.researchgate.net/publication/283497019_Reablement_in_community-dwelling_older_adults_a_randomised_controlled_trial
- See also: Published cost-effectiveness study — http://healtheconomicsreview.springeropen.com/articles/10.1186/s13561-016-0092-8